CLINICAL TRIAL: NCT02939729
Title: The Effect of a Physiotherapy Prehabilitation Programme on Postoperative Outcomes in Patients Undergoing Cardiac or Thoracic Surgery
Brief Title: Physiotherapy Prehabilitation in Patients Undergoing Cardiac or Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16/CARD/18
Record Dates: First submitted 2016-08-25; First posted 2016-10-20 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease; Lung Cancer; Lung Tumor
Keywords: prehabilitation; physiotherapy; cardiac; thoracic; preoperative
MeSH Terms: conditions — Coronary Artery Disease; Lung Neoplasms | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Experimental): This group will receive standard preoperative information and education and be provided with a physiotherapy prehabilitation programme. This programme will be carried out from time of consenting to participate in the study until day of admission to surgery for cardiac or thoracic surgery. The prehabilitation programme consists of: walking programme, deep breathing exercises and tidal volume measurement using the incentive spirometer.
  Interventions: Other: Walking Programme; Device: Incentive Spirometer; Other: Deep Breathing Exercises
- Standard Care (No Intervention): This group will receive standard preoperative information and education only.

INTERVENTIONS:
Other: Walking Programme — Walking programme measured by daily step count on pedometer provided to participant. Participants will be advised to increase daily step count from their baseline measure - realistic incremental rise according to individual ability and symptoms. Daily step count will be recorded in a participant study diary.
  Arms: Prehabilitation
Device: Incentive Spirometer — An incentive spirometer is a device used to measure lung tidal volumes. Participants will be asked to use the incentive spirometer to measure their tidal volume daily. Participants will record daily tidal volume measurement in the participant diary. A physiotherapist will teach participants how to use the incentive spirometer and provide an instruction sheet.
  Arms: Prehabilitation
Other: Deep Breathing Exercises — Participants will be taught deep breathing exercises - these are the same deep breathing exercises shown to all patients after cardiac surgery as part of chest physiotherapy treatment. Participants will be asked to carry out deep breathing exercises at home during the prehabilitation phase. An instruction sheet for the deep breathing exercises will be provided to participants.
  Other Names: Breathing Exercises
  Arms: Prehabilitation

SUMMARY:
The purpose of this study is to determine the effects of a physiotherapy prehabilitation programme (walking and deep breathing exercises) in cardiac or thoracic patients by measuring changes in lung volumes, functional capacity physiotherapy length of stay postoperatively.

DETAILED DESCRIPTION:
Preoperative rehabilitation or "Prehabilitation" can be defined as "the process of enhancing the functional capacity of the individual to enable him or her to withstand a stressful event". Prehabilitation is a relatively new concept with emerging evidence demonstrating a reduction in length of hospital stay and disability, improved functional capacity and quality of life as well as fewer peri-operative complications compared to usual care.

Patients who are awaiting Cardiothoracic surgery are often fearful of being physically active, however extended periods of physical inactivity lead to a loss of muscle mass, physical deconditioning and pulmonary complications which can in turn lead to decreased quality of life, higher levels of morbidity, increased hospital length of stay and even fatality.

Based on literature supporting the positive effects of physical activity, physiotherapy prehabilitation aims to enhance functional exercise capacity in patients undergoing Cardiothoracic surgery and hence minimising the risk of postoperative morbidity and enhancing postsurgical recovery. Although there is evidence for prehabilitation in cardiothoracic specialties these are mainly within heart failure patients therefore not comparable to patients undergoing CABG or lobectomy surgeries.

The aim of this study is to determine whether a home based preoperative prehabilitation programme improves patients' functional capacity, as measured by a 6 minute walk test (6MWT) prior to surgery and improve post surgical recovery and recovery of functional capacity earlier. This study will compare functional capacity levels from baseline (at time of being accepted for surgery) and on the day of admission for surgery. Secondary aims are to determine functional capacity prior to discharge from hospital and at 6-8 week follow up appointment. Increasing maximal tidal volumes preoperatively would in turn decrease the chance of atelectasis postoperatively thereby decreasing pulmonary complications. Time to achieve discharge criteria from physiotherapy and total post-operative hospital length of stay will be assessed. Patient health related satisfaction will be assessed using the EQ-5D. The endpoint of this study will be when the patient returns for their routine 6-8 week follow up appointment and completes final 6MWT, tidal volume (TV) measurement and EQ-5D.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery -

  * Patients undergoing primary CABG surgery
  * Age >18 years old
  * Able to mobilise independently with/without a walking aid

Thoracic surgery -

* Patients undergoing lobectomy surgery
* Age >18 years old
* Able to mobilise independently with/without a walking aid

Exclusion Criteria:

* Cardiac surgery -

  * Unstable angina (Grade IIIb as described in Braunwald Classification of Unstable Angina/ angina at rest within the last 48 hours)
  * History of cerebrovascular accident (CVA)
  * History of traumatic brain injury (TBI)
  * Patients who require interpreter
  * Falls risk as classified by the GJNH falls risk document
  * Patients included within cardiac surgery ERAS programme
  * Any patient who lacks capacity to consent
  * Patients who are admitted for urgent or emergency cardiac surgery e.g. aortic stenosis

Thoracic surgery -

* Unstable angina (Grade IIIb as described in Braunwald Classification of Unstable Angina/ angina at rest within the last 48 hours)
* History of cerebrovascular accident (CVA)
* History of traumatic brain injury (TBI)
* Patients who require interpreter
* Falls risk as classified by the GJNH falls risk document
* Any patient who lacks capacity to consent
* Patients who are admitted for urgent or emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Difference between groups functional activity from baseline to point of admission for surgery as measured by the 6MWT. | From date of randomisation to date of admission for surgery (up to 8 weeks)
  The 6MWT is a validated test that requires no exercise equipment or "advanced" training for the assessor. Walking is an activity carried out on a daily basis by most people. The 6MWT measures the distance that a person can walk on a flat surface over a period of 6 minutes. The majority of activities of daily living are carried out at "sub-maximal" levels similar to the level of exertion of the 6MWT as the patient sets their own intensity (American Thoracic Society 2002). A review of functional walking tests suggested that "the 6MWT is easy to administer, better tolerated, and more reflective of activities of daily living than the other walk tests" (Solway et al 2001). Other prehabilitation studies have used the 6MWT as an outcome measure of functional activity therefore is widely accepted as a reliable measure of functional activity (Sawatzky et al 2014; Carli et al 2010; Gillis et al 2014).

SECONDARY OUTCOMES:
Functional capacity as measured by 6MWT on day of discharge and at return clinic appointment (up to 8 weeks) | Date of discharge from physiotherapy and at return clinic appointment (up to 8 weeks)
  Measure of level of physical activity measured in metres
Tidal Volume (TV) measures with incentive spirometer. | At baseline, preoperative, postoperative days 1, 2 and 3 and at return clinic appointment (up to 8 weeks)
  Lung volume measure in mls
Day of discharge from Physiotherapy. | Once all physiotherapy criteria have been met (approximately 3 to 5 days).
  Physiotherapy discharge criteria: mobilising safely and independently with or without walking aid approximately 100 metres; independently managing chest and safely completed stairs assessment (approximately post op day 3 to 5).
Total postoperative hospital length of stay. | Once all hospital discharge criteria have been met (approximately 5-7 days).
  Total post operative hospital length is days in hospital after surgery.
EQ-5D score. | At baseline and follow up clinic appointment (up to 8 weeks).
  A standardized and validated measure of health status which can be used in a wide range of health conditions. It is a simple method which patients can complete at the beginning and end of treatment. It encompasses five dimensions of health: mobility, ability to self care, ability to complete activities of daily living, pain and discomfort, and anxiety and depression (Chartered Society of Physiotherapists, 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Nolan, Grad Dip, Study Chair — National Waiting Times Centre Board; Katie L Lyon, MSc, Principal Investigator — National Waiting Times Centre Board
Locations (1):
- Golden Jubilee National Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ditmyer MM, Topp R, Pifer M. Prehabilitation in preparation for orthopaedic surgery. Orthop Nurs. 2002 Sep-Oct;21(5):43-51; quiz 52-4. doi: 10.1097/00006416-200209000-00008. PMID 12432699
- [Background] Topp R, Ditmyer M, King K, Doherty K, Hornyak J 3rd. The effect of bed rest and potential of prehabilitation on patients in the intensive care unit. AACN Clin Issues. 2002 May;13(2):263-76. doi: 10.1097/00044067-200205000-00011. PMID 12011598
- [Background] Santa Mina D, Clarke H, Ritvo P, Leung YW, Matthew AG, Katz J, Trachtenberg J, Alibhai SM. Effect of total-body prehabilitation on postoperative outcomes: a systematic review and meta-analysis. Physiotherapy. 2014 Sep;100(3):196-207. doi: 10.1016/j.physio.2013.08.008. Epub 2013 Nov 13. PMID 24439570
- [Background] Carli F, Charlebois P, Stein B, Feldman L, Zavorsky G, Kim DJ, Scott S, Mayo NE. Randomized clinical trial of prehabilitation in colorectal surgery. Br J Surg. 2010 Aug;97(8):1187-97. doi: 10.1002/bjs.7102. PMID 20602503
- [Background] Mooney M, Fitzsimons D, Richardson G. "No more couch-potato!" Patients' experiences of a pre-operative programme of cardiac rehabilitation for those awaiting coronary artery bypass surgery. Eur J Cardiovasc Nurs. 2007 Mar;6(1):77-83. doi: 10.1016/j.ejcnurse.2006.05.002. Epub 2006 Jul 10. PMID 16831570
- [Background] Valkenet K, van de Port IG, Dronkers JJ, de Vries WR, Lindeman E, Backx FJ. The effects of preoperative exercise therapy on postoperative outcome: a systematic review. Clin Rehabil. 2011 Feb;25(2):99-111. doi: 10.1177/0269215510380830. Epub 2010 Nov 8. PMID 21059667
- [Background] Carli F, Zavorsky GS. Optimizing functional exercise capacity in the elderly surgical population. Curr Opin Clin Nutr Metab Care. 2005 Jan;8(1):23-32. doi: 10.1097/00075197-200501000-00005. PMID 15585997
- [Background] McKelvie RS, Teo KK, Roberts R, McCartney N, Humen D, Montague T, Hendrican K, Yusuf S. Effects of exercise training in patients with heart failure: the Exercise Rehabilitation Trial (EXERT). Am Heart J. 2002 Jul;144(1):23-30. doi: 10.1067/mhj.2002.123310. PMID 12094184
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Solway S, Brooks D, Lacasse Y, Thomas S. A qualitative systematic overview of the measurement properties of functional walk tests used in the cardiorespiratory domain. Chest. 2001 Jan;119(1):256-70. doi: 10.1378/chest.119.1.256. PMID 11157613
- [Background] Sawatzky JA, Kehler DS, Ready AE, Lerner N, Boreskie S, Lamont D, Luchik D, Arora RC, Duhamel TA. Prehabilitation program for elective coronary artery bypass graft surgery patients: a pilot randomized controlled study. Clin Rehabil. 2014 Jul;28(7):648-57. doi: 10.1177/0269215513516475. Epub 2014 Jan 23. PMID 24459173
- [Background] Gillis C, Li C, Lee L, Awasthi R, Augustin B, Gamsa A, Liberman AS, Stein B, Charlebois P, Feldman LS, Carli F. Prehabilitation versus rehabilitation: a randomized control trial in patients undergoing colorectal resection for cancer. Anesthesiology. 2014 Nov;121(5):937-47. doi: 10.1097/ALN.0000000000000393. PMID 25076007